CLINICAL TRIAL: NCT02061475
Title: The Efficacy and Safety of Lidocaine Patches for Attenuating the Pain of Venipuncture Intravenous Cannulation Before Surgery: a Multicenter, Randomized, Double -Blind, Placebo-controled and Parallel-group Designed Clinical Trail
Brief Title: Lidocaine Patches for Attenuating the Pain of Venipuncture Intravenous Cannulation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Nitto Denko Corporation (Industry); Giant Med-Pharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LCLDKY-13115
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-06

CONDITIONS: We Focus on the Pain of Venipuncture and Intravenous Cannulation
Keywords: Lidocaine patches; Pain; Intravenous cannulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine Patches (Active Comparator)
  Interventions: Drug: Lidocaine Patches
- Placebo Patches (Placebo Comparator)

INTERVENTIONS:
Drug: Lidocaine Patches
  Arms: Lidocaine Patches

SUMMARY:
Venipuncture and intravenous cannulation are the most common painful procedures, especially for the penitents who must receive large diameter venous catheter before surgery. In present study we would evaluate the safety and validity of lidocaine patches releasing such pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who want to participate present study and sign the informed consent form
* Age from 18 to 65 years old
* Patients who need intravenous cannulation before surgery
* ASA class I-II and selected patients

Exclusion Criteria:

* Allergic to lidocaine or any other amide local anesthetics or any other medicine
* Allergic skin(allergic to past agent or other topical used medicine)
* Skin injured or inflection exist in the local site to patch
* Sensation disturbed in any limb
* Severe liver and kidney original disease:blood Aspertate aminotransferase and Alanine transaminase increased 1.5 times more than normal concentration; blood creatinine is higher than the normal range.
* Hemoglobin <80g/L
* ECG is significantly abnormal
* pregnant or possible pregnant or breastfeeding woman
* Patient who has consciousness disturbance can not make credible dialog with investigator.
* Those who are using other medicine may affect the evaluation of present patch
* Those who have participated in other clinical trail in the past three months
* Those excluded by investigator believed other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The efficiency of lidocaine patches for attenuating the pain of venipuncture intravenous cannulation before surgery | Two minters after intravenous cannulation
  VAS score will be evaluated two minters after intravenous cannulation in both group with lidocaine patches or not.
Skin response after intravenous cannulation | Thirty minters after intravenous cannulation
  Local skin response to the lidocaine patches will be evaluated thirty minters after intravenous cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Xiangrui Wang, Dr., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Yanhua Zhao, Dr., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guanzhou First people's Hospital, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changhai, Hunan
  - The First Affiliate Hospital of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital Affiliated to Shanghai Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality